CLINICAL TRIAL: NCT07211347
Title: Percutaneous Blockade Protocol of the Stellate Ganglion in Patients With Refractory Electrical Storm
Brief Title: Percutaneous Blockade of the Stellate Ganglion in Electrical Storm
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7.441.184
Record Dates: First submitted 2025-08-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Electrical Storm; Stellate Ganglion Block; Ventricular Arrhythmia
Keywords: Ventricular Arrhythmia; Electrical Storm; Stellate ganglion block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block (Active Comparator)
  Interventions: Procedure: Stellate Ganglion Block
- Standard Treatment (No Intervention)

INTERVENTIONS:
Procedure: Stellate Ganglion Block — There is no randomized clinical study in the literature that evaluated the efficacy and safety of the stellate ganglion infiltration procedure in patients with electrical storm.
  Arms: Stellate Ganglion Block

SUMMARY:
There is no randomized clinical study in the literature that evaluated the efficacy and safety of the stellate ganglion infiltration procedure in patients with electrical storm. So far, case reports and retrospective studies suggest that such a strategy should be considered in cases refractory to initial therapy. In this scenario, the European and American guidelines for the treatment of ventricular arrhythmias recommend autonomic modulation in this setting, but only with a level of recommendation IIb (1,2). This project aims to evaluate the effect of stellate ganglion infiltration in patients with electric storm refractory to initial clinical measures. It is a randomized clinical trial where patients will receive treatment with a lidocaine and bupivacaine anesthetic solution or no intervention. The effect of the intervention will be considered positive when there is a reduction of arrhythmic events of at least 50% in the 12 hours immediately after.

DETAILED DESCRIPTION:
The study aims to evaluate the reduction of arrhythmic events following stellate ganglion blockade in patients with electrical storm refractory to initial clinical measures.

Hypothesis Stellate ganglion infiltration is an effective neuromodulation strategy for controlling arrhythmic events in patients with electrical storm awaiting definitive therapy.

Methodology This is a single-center randomized study investigating the efficacy of stellate ganglion blockade in patients with electrical storm refractory to initial clinical measures.

Participant Selection and Sample Size Participants will include patients admitted to the Emergency Unit or any Intensive Care Unit with a diagnosis of refractory electrical storm. Based on the STAR study, which reported a median of 6 arrhythmic events before SGB (IQR: 3 to 15.8), and aiming for at least a 50% reduction in arrhythmias in the active group post-procedure (with no expected change in the placebo group), a sample size of 32 patients per group was calculated (alpha = 0.05, power = 80%, two-tailed test).

Definitions Electrical storm (ES) is defined as three or more episodes of ventricular arrhythmias (including appropriate ICD therapies), separated by at least 5 minutes, within 24 hours. Refractory ES is defined as recurrent arrhythmias despite antiarrhythmic drug administration. Patients requiring discontinuation of antiarrhythmics due to adverse events will also be eligible for SGB. An arrhythmic event is defined as an episode of sustained VT or VF (>30 seconds or unstable), treated or not with antitachycardia pacing (ATP), electrical therapy, ICD shock, or external defibrillation. Pre-specified complications include: simple hematoma, hematoma requiring intervention, symptoms due to anesthetic absorption, brachial plexus injury, simple vascular injury, and vascular injury requiring intervention.

Randomization Randomization will be performed by a medical professional not involved in the infiltration procedure and blinded to data analysis, using the "Randomizer for Clinical Trial" software.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with structural heart disease and a diagnosis of refractory electrical storm, or those who require discontinuation of antiarrhythmics due to adverse events or contraindications to standard therapy.

Exclusion Criteria:

* Patients under 18
* History of heart transplant or prior cardiac denervation surgery
* Anatomical contraindications for the procedure (prior neck surgery, burns, large scars, or thyroid goiter).
* Genetically related polymorphic VT
* End-stage renal disease on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in arrhythmic events | 12 hours immediately after the blockade compared to the 12 hours immediately before
  A ≥50% reduction in arrhythmic events (VT/VF)

SECONDARY OUTCOMES:
ICD therapies | 12 hours immediately after stellate ganglion block (SGB) compared to the 12 hours immediately before
  Reduction in the number of ATPs/ICD shocks
Urgent ablation and other invasive therapies | 72 hours after the blockade
  urgent ablation and other invasive therapies (e.g., intra-aortic balloon pump placement or intubation for deep sedation)

CONTACTS AND LOCATIONS:
Overall Officials: Maurício I Scanavacca, MD, PhD, Principal Investigator — Instituto do Coração - HC/FMUSP
Locations (1):
- Clinical Research Center of the Heart Institute - University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savastano S, Baldi E, Compagnoni S, Rordorf R, Sanzo A, Gentile FR, Dusi V, Frea S, Gravinese C, Cauti FM, Iannopollo G, De Sensi F, Gandolfi E, Frigerio L, Crea P, Zagari D, Casula M, Sangiorgi G, Persampieri S, Dell'Era G, Patti G, Colombo C, Mugnai G, Notaristefano F, Barengo A, Falcetti R, Perego GB, D'Angelo G, Tanese N, Currao A, Sgromo V, De Ferrari GM; STAR study group. Electrical storm treatment by percutaneous stellate ganglion block: the STAR study. Eur Heart J. 2024 Mar 7;45(10):823-833. doi: 10.1093/eurheartj/ehae021. PMID 38289867